CLINICAL TRIAL: NCT00031018
Title: Prevention of Cognitive Decline in Alzheimer's Disease by Ingested Interferon Alpha
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR02558-0120
Record Dates: First submitted 2002-02-20; First posted 2002-02-22 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Memory Disorders; Alzheimer's Disease
Keywords: Inflammation; immunosenescence; autoimmunity; atherosclerosis; pro-inflammatory cytokines; Hayflick phenomenon
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease; Inflammation; Autoimmune Diseases; Atherosclerosis | interventions — Donepezil; Interferon alpha-2

INTERVENTIONS:
Drug: Aricept
Drug: IFN-alpha2A

SUMMARY:
In this phase I-II parallel design, randomized, double-blind clinical trial we will determine if 3,000 or 30,000 units ingested hrIFN-a prevents deterioration of cognitive functioning in patients with dementia of Alzheimer's type (AD) and whether ingested hrIFN-a treatment decreases acute phase reactants and pro-inflammatory cytokine IL-6 in mild to moderate AD. We predict that the novel anti-inflammatory agent ingested human recombinant interferon alpha (hrIFN-a) will modulate inflammation and inhibit the natural history of AD progression. If you are eligible, you will receive Aricept for 5 weeks (donezepil) and thereafter in addition to Aricept either placebo (inactive substance) or interferon alpha at 3,000 or 30,000 units every day for 12 months.

DETAILED DESCRIPTION:
Inflammatory mechanisms contribute to neurodegeneration in AD. Acute phase proteins such as the antichymotrypsin (a1ACT), pro-inflammatory cytokines IL-6 and IL-1, and activated microglial cells are all associated with neuritic plaques. a1ACT levels are elevated in AD, correlate with cognitive decline and serve as a biological marker of intervention. a1ACT is intimately associated with the 42-AA b peptide (Ab) in filamentous amyloid deposits and stimulates the polymerization of Ab into amyloid filaments. IL-6 is found in AD cortices prior to the onset of neuritic change, serum and stimulated PMNC IL-6 levels are higher in AD, and may induce b-amyloid protein deposition. Microglia, CNS resident inflammatory cells, produce IL-6 within the adult human brain, are IL-1a +, and are a prominent component of the neuritic plaque. Because the pathogenesis of AD appears in part immune mediated, we propose testing directly in humans whether ingested IFN-a can ameliorate AD. Because there is no good model for inflammation in animal models of AD, we will directly determine in humans 1) if 3,000 or 30,000 IU hrIFN-a inhibits the natural history rate of cognitive decline in mild to moderate AD using neuropsychological instruments as primary and secondary outcome measures that 2) correlates with inhibition of acute phase reactants and pro-inflammatory IL-6. If this novel anti-inflammatory agent inhibits the natural history rate of cognitive decline in AD in this pilot phase II trial, this would provide the preliminary data to submit a phase III clinical trial.

IFNs administered by the oral route show a systemic effect. Oral IFN-a caused neutropenia in mice. In contrast to their i.p. administration, oral IFN-a did not result in the presence of detectable levels of IFNs in the blood. Circulating specific antibody to IFN blocked the neutropenic effects of i.p. IFN, but did not block the neutropenic effects of the oral IFNs (2). Therefore, we examined the expression of antiviral MxA message, a type 1 IFN-specific induced signal, as a sensitive marker for type 1 IFN interaction with lymphoid cells in the gut-associated lymphoid tissue (GALT) using semi-quantitative RT-PCR on splenocytes from mice and PMNC from man after IFN-a ingestion. Both mice and man demonstrated inducible levels of Mx mRNA after ingesting IFN-a. Murine spleen T cells and CD8+ T cells also demonstrated upregulation of Mx mRNA. Therefore, ingested IFN-a acts via established pathways of type 1 IFN signalling (3). Elevated levels of activated T cells, mainly of the CD8+ (cytotoxic/suppressor) phenotype, are found in AD brains in contact with microglial cells (4). Interestingly, peripheral CD8+ T cells are depleted in AD patients (5). Lymphocytes bearing T helper and T cytotoxic/suppressor cell antigens are found in hippocampus and temporal cortex in AD (6,7). The data above suggest that lymphocytes are part of inflammation in AD, and potential immunomodulatory T and CD8+ T cells that contact ingested non-absorbed IFN in the GALT could migrate to the brain and decrease inflammation.

ELIGIBILITY:
Inclusion Criteria:

Males and females, age 50 or greater. Possible or probable dementia of the Alzheimer Type defined by NINDS-ARDA criteria with dementia of at least one year duration.

Folstein MMSE Score 10-24 inclusive. Vision, hearing, speech, motor function and comprehension must be adequate for compliance with all testing procedures.

Exclusion Criteria:

Absence of a reliable caregiver. Clinical or radiological evidence for other neurological disorders such as Parkinson's disease, normal pressure hydrocephalus, multi-infarct dementia, idiopathic seizure disorder, CNS infectious disease.

History of major psychiatric disorders; schizophrenia and unipolar or bipolar depression.

Presence of any significant medical disorder which might cause or contribute to dementia such as B12 or folic acid deficiency, untreated hypothyroidism, history of significant alcohol abuse (within the past 10 years).

Patients with recent (< 2 years) hematologic/oncologic disorders (other than basal or squamous cell carcinoma of the skin.

Patients with recent (< 3 months) myocardial infarction, poorly controlled CHF, surgery for peripheral vascular disease, or coronary artery bypass surgery.

Evidence of clinically significant or unstable active GI, hepatic or pulmonary disease.

History of documented stroke or more than one confirmed TIA. Any condition which would make the patient or caregiver, in the opinion of the principal investigator unsuitable for the study.

Patients with known hypersensitivity to Donezepil HCL or other piperidine containing drugs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas - Houston, Gerontology Center of the UTMSI, Houston, Texas, United States

REFERENCES:
- [Background] Brod SA. Unregulated inflammation shortens human functional longevity. Inflamm Res. 2000 Nov;49(11):561-70. doi: 10.1007/s000110050632. PMID 11131295